CLINICAL TRIAL: NCT00641823
Title: Objective Functional Outcome Measures in Orthopedic Surgery Using Advanced Tracking Technologies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Yair Barzilay, Hadassah Medical Organization
Other Study IDs: BARZ-002HMO-CTIL
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Orthopedic Disorders
Keywords: Orthopedic Surgical Procedures
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- 1
- 2
- 3

SUMMARY:
The proposed project will address the measurement and ramifications of out-of-home mobility problems in various orthopedic disorders in an innovative way, using advanced tracking technologies.

ELIGIBILITY:
Inclusion Criteria:

* Unwillingness to sign informed consent.

Exclusion Criteria:

* Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from osteoarthritis of the hips and knees, patient suffering from spinal claudication, and unimpaired controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2015-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel